CLINICAL TRIAL: NCT06457230
Title: Exploration of the Intervention Mechanism and Efficacy of Paired-pulse rTMS Treatment for Methamphetamine Use Disorder Based on the mPFC-Cerebellum
Brief Title: Paired-pulse rTMS Treatment for Methamphetamine Use Disorder Based on the mPFC-Cerebellum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Hanyang Drug Rehabilitation Center (Unknown); Chengdu Drug Rehabilitation Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MZhao-015
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Methamphetamine Use Disorder
Keywords: Repetitive transcranial magnetic stimulation; Cerebellum; Frontopolar cortex; Methamphetamine; Cortico-Cortical Paired Associative Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Cerebellar Stimulation + Sham mPFC Stimulation Group (Sham Comparator): This is the sham stimulation group. The coil will be placed vertically over the cerebellar and mPFC brain regions, allowing participants to perceive the coil's vibration and sound without receiving effective intervention. All other stimulation parameters are identical to those in the active intervention group.
  Interventions: Device: Sham Intervention Group
- Cerebellar-mPFC Dual-Coil Paired-Pulse TMS Intervention Group (Experimental): The stimulation protocol involved delivering a pulse to the cerebellum first, followed by a pulse to the mPFC after a 6ms inter-stimulus interval (ISI). This 6ms interval was determined based on findings from our prior mechanistic study.
  Interventions: Device: Paired Associative Stimulation Targeting the Cerebellar-mPFC

INTERVENTIONS:
Device: Paired Associative Stimulation Targeting the Cerebellar-mPFC — The protocol consisted of 180 pulse trains. Each train contained 5 pulse pairs delivered over 1 second, resulting in a stimulation frequency of 5 Hz. Within each pulse pair, the cerebellum was stimulated first, followed by the mPFC after a 6-ms inter-stimulus interval (ISI). In total, 900 pulse pairs were administered, and a complete intervention session lasted 11 minutes and 57 seconds.
  Arms: Cerebellar-mPFC Dual-Coil Paired-Pulse TMS Intervention Group
Device: Sham Intervention Group — The coil will be placed vertically over the cerebellar and mPFC brain regions, allowing participants to perceive the coil's vibration and sound without receiving effective intervention. All other stimulation parameters are identical to those in the active intervention group.
  Arms: Sham Cerebellar Stimulation + Sham mPFC Stimulation Group

SUMMARY:
To investigate the mechanism and efficacy of a novel repetitive transcranial magnetic stimulation (rTMS) intervention model with paired medial prefrontal cortex (mPFC) -cerebellar pulses on methamphetamine use in patients and to develop a novel physiotherapeutic intervention to optimise the treatment and management of addicted patients.

DETAILED DESCRIPTION:
Numerous studies have shown that impaired mPFC-cerebellar functional connectivity leads to impaired social preferences and behavioural flexibility and more persistent drug use in addicts. Cerebellar and mPFC paired-pulse rTMS interventions may enhance functional connectivity, effectively modulate cerebellar-prefrontal loops, reduce craving, improve cognitive flexibility, and reduce relapse risk. The aim of this project is to investigate the mechanism and efficacy of a novel paired-pulse rTMS intervention targeting the mPFC-cerebellar circuit in patients with methamphetamine use disorder, in order to develop innovative physiotherapeutic interventions and to optimize treatment and clinical management for individuals with addiction.

Prior to initiating the intervention, it was essential to determine the optimal inter-stimulus interval (ISI) for the cerebellar-mPFC paired associative stimulation. Therefore, a mechanistic study was conducted from December 2024 to June 2025 at the Chengdu Drug Rehabilitation Center in Sichuan Province before the interventional trial commenced. A mixed design was employed, contrasting single-pulse mPFC stimulation with cerebellum→mPFC cortico-cortical paired associative stimulation (ccPAS) at inter-stimulus intervals of 6 ms and 45 ms. The results revealed that individuals with methamphetamine use disorder exhibited aberrant cerebellar-mPFC circuit connectivity compared to healthy controls. Importantly, cerebellar-mPFC ccPAS with a 6-ms ISI was found to specifically modulate this inter-regional circuit dysfunction.

Therefore, based on the identified 6-ms cerebellar-mPFC stimulation interval, the current interventional study continues to implement a long-term, dual-coil combined stimulation protocol to further evaluate and establish its therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria

1. Primary substance of abuse is methamphetamine.
2. Meets the DSM-5 diagnostic criteria for severe methamphetamine use disorder (≥6 symptoms present within the past year).
3. Age: 18-60 years.
4. Education level of primary school or above, with the ability to comprehend questionnaires and behavioral tasks.
5. Normal vision and hearing; right-handed.
6. No prior participation in any TMS-related intervention therapy.

Exclusion Criteria

1. Presence of any metallic implants (e.g., dental prostheses, orthodontic braces, bone fixation plates, aneurysm clips, intrauterine devices) or implanted medical devices such as cardiac pacemakers or neurostimulators.
2. Chronic or severe somatic diseases (e.g., cardiac conditions, uncontrolled hypertension, physical disabilities).
3. Comorbid psychiatric disorders (e.g., schizophrenia, depressive disorders, anxiety disorders).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
cognitive flexibility | Probabilistic reversal learning task: baseline, post-intervention, and at a follow-up session one weeks later; Volatile reversal learning task and Wisconsin Card Sorting Test: baseline and post-intervention; The CFI scale: baseline.
  Based on tasks and scales assessing cognitive flexibility, including: 1.Probabilistic reversal learning task (The matching of symbols and pictures was reversed without informing the subjects and their cognitive flexibility in the reversed condition was assessed); 2.Volatile reversal learning task (participants were presented with two stimuli associated with their potential feedback magnitude. They were instructed to choose one of the two stimuli to receive feedback, but only one stimulus would result in feedback. ); 3.The Wisconsin Card Sorting Test (WCST) (a classic neuropsychological task where participants match response cards to four key cards based on hidden sorting rules (color, shape, or number). They receive "right" or "wrong" feedback after each match and must deduce the current rule, which changes without warning after several consecutive correct matches.); 4. The Cognitive Flexibility Inventory (CFI) scale is a 20-item self-report measure.

SECONDARY OUTCOMES:
Craving | before the intervention (baseline), immediately after the intervention (post-intervention), and at a follow-up session one weeks later.
  1、The intensity of psychological craving in MA dependents was assessed using the Visual Analogue Scale (VAS), where individuals rated their cravings on a scale from 0 to 100, with higher scores indicating greater levels of craving. 2、Desires for drug questionnaire (DDQ) consists of 13 items designed to assess an individual's current thoughts and preoccupations related to drug use. 3、Obsessive Compulsive Drug Use Scale (OCDUS)consists of 13 items designed to assess an individual's current thoughts and preoccupations related to drug use.
Electroencephalographic (EEG) Electrophysiological Results | before the intervention (baseline), immediately after the intervention (post-intervention), and at a follow-up session one weeks later.
  This includes analyses of TMS-EEG, resting-state EEG, and task-state EEG data across temporal, frequency, and time-frequency domains.
response inhibition | SST task: baseline, post-intervention, and at a follow-up session one weeks later; BIS-11 scale: baseline.
  The Stop-Signal Task (SST) is a seminal experimental paradigm in cognitive psychology and neuroscience designed to objectively measure an individual's response inhibition-the ability to actively suppress a prepotent or already-initiated motor response. To gain a more comprehensive understanding of an individual's inhibitory control, it is highly informative to complement this with a trait-based, self-reported measure of impulsivity. The Barratt Impulsiveness Scale, Version 11 (BIS-11) serves this purpose. The BIS-11 is a widely validated questionnaire that assesses stable, cross-situational personality traits related to impulsivity across three core dimensions: Attentional Impulsiveness (inability to focus attention), Motor Impulsiveness (tendency to act without thinking), and Non-Planning Impulsiveness (lack of forethought).
Depression | before the intervention (baseline), immediately after the intervention (post-intervention), and at a follow-up session one weeks later.
  The reduction rate of Beck Depression Inventory (BDI) scores was calculated from baseline to post-intervention and follow-up assessments to quantify the decrease in depressive symptom severity.
Anxiety | before the intervention (baseline), immediately after the intervention (post-intervention), and at a follow-up session one weeks later.
  The reduction rate in the Beck Anxiety Inventory (BAI) scores was calculated from baseline to post-intervention and follow-up assessments to quantify the decrease in anxiety symptom severity.
stress levels | before the intervention (baseline), immediately after the intervention (post-intervention), and at a follow-up session one weeks later.
  The reduction rate of Perceived Stress Scale (PSS) scores was calculated from baseline to post-intervention and follow-up assessments to quantify the decrease in perceived stress levels.
sleep quality | before the intervention (baseline), immediately after the intervention (post-intervention), and at a follow-up session one weeks later.
  The reduction rate of Pittsburgh Sleep Quality Index (PSQI) global scores was calculated from baseline to post-intervention and follow-up assessments to quantify the improvement in sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, PhD, Study Chair — Shanghai Mental Health Center
Locations (1):
- Min Zhao, PhD, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification, will be made available at the discretion of the corresponding author, following a formal request and execution of a data use agreement.
Supporting Information: Study Protocol, SAP, ICF